CLINICAL TRIAL: NCT04758026
Title: Survivorship and Late Effects in Head and Neck Cancer Survivors
Brief Title: H&N Cancer; Survivorship and Late Effects
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Cecilie Delphin Amdal, Senior Oncologist, PhD, Researchgroupleader skin and head and neck cancer, Department of Oncology, Oslo University Hospital
Other Study IDs: 2018-21
Record Dates: First submitted 2021-02-04; First posted 2021-02-17 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Neoplasms; Survivorship
Keywords: Patient Reported Outcome Measure; Quality of Life; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample With biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study on late effects after modern treatment in long-term survivors of head and neck cancer (HNC). Participants fill in questionnaires and participate at a one day visit at the hospital including blood sample with biomarkers, clinical examination, audiometry, oral radiological examination and oral examination. Data on patients' medical history collected from medical records including radiology images and digital radiotherapy plans.This will allow adjustments of treatment planning and improved treatment decisions for patients at risk, and improve information and follow up for future patients.

DETAILED DESCRIPTION:
The purpose of this study is to provide knowledge on late effects and mortality risk after modern treatment in long-term survivors of head and neck cancer (HNC). This will allow adjustments of treatment planning and improved treatment decisions for patients at risk, and improve information and follow up for future patients. For head and neck cancer (HNC) survivors of today, with the rising proportion of HPV induced cancer and with improved modern treatment, the late effects and mortality risk has changed compared to survivors previous decades.

The investigators will assess the prevalence and severity of a broad range of late effects and identify associated risk factors for the following late effects;

* Chronic fatigue
* Hearing loss and tinnitus
* Oral late effects, including taste and smell disturbances and osteoradionecrosis
* Dysphagia and malnutrition
* Body image, intimacy and endocrine dysfunction

In addition,possible biological explanatory mechanisms for fatigue and possibly other selected late effects will be explored. Data will be compared to age and gender matched reference data for those where this is available.

Design: a cross-sectional study

Assessments: Patient-reported questionnaires, blood sample with biomarkers, clinical examination, audiometry, oral radiological examination and oral examination. Data on patients' medical history collected from medical records including radiology images and digital radiotherapy plans.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically verified invasive carcinoma of the head and neck region; ICD10: C01, C02.0 - C02.9; C03.0 - C03.9; C04.0 - C04.9; C05.0 - C05.9; C06.0 - C06.9; C07; C08.0 - C08.9; C09.0 - C09.9; C10.0 - C10.9; C11.0 - C11.9; C12; C13.0 - C13.9; C14.0 - C14.9; C30; C31.0 - C31.9; C32.0 - C32.9, C77.0
* Diagnosed 2006- 2012
* Ability to understand and respond to the questionnaires
* Ability to attend the clinical examination
* Informed consent received

Exclusion Criteria:

* Unwillingness to answer HRQL questionnaires
* Patients under ongoing treatment for secondary cancer or relapse at the time of the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HNC survivors treated at OUH in the period from 2006 to 2012 are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of late effects after head and neck cancer treatment measured with patient-reported questionnaires | June 2022
  Assess prevalence of fatigue, dysphagia, xerostomia, hearing problems, oral health, body image and intimacy in surivors of head and neck cancer more than 5 years after treatment. Patients filled in a set of patient-reported questionnaires: 1) EORTC core quality of life questionnaire, the EORTC QLQ-C30 version 3, 2) EORTC disease specific module, the EORTC QLQ-H&N35 3) The Fatigue Questionnaire, 4) The scale for chemotherapy induced neurotoxicity (SCIN), 5) EORTC-QLQ-OH15, 6) Body image scale.

SECONDARY OUTCOMES:
Risk factors for late effects after head and neck cancer treatement | June 2022
  to explore associated risk factors for fatigue, dysphagia, xerostomia, hearing problems, oral health in surivors of head and neck cancer more than 5 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data from 50-100 of the participants will be included in the EORTC 1629 - Late toxicity and long-term quality of life in head and neck cancer survivors
Supporting Information: Study Protocol, CSR
Time Frame: 2020